CLINICAL TRIAL: NCT06122922
Title: Xenon MRI in Stable Patients With Pulmonary Hypertension
Brief Title: Xenon MRI in Stable Pulmonary Hypertension (Jupiter AUGEAN)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Bastiaan Driehuys (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, IND Holder, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00113235
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Stable Pulmonary Arterial Hypertension (Other): Stable on current treatment regimen and not planning to undergo initiation of new therapy for at least 3 months Intervention: Drug: 129Xe Hyperpolarized
  Interventions: Drug: Hyperpolarized Xe129

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Hyperpolarized Xenon Gas

SUMMARY:
The objective of this project is to determine how pulmonary vascular remodeling in Pulmonary Arterial Hypertension (PAH) at cellular and pathological level is associated with gas exchange physiology changes and hemodynamics (monitored with 129Xe MRI/MRS) and how these signals change with disease progression or treatment.

DETAILED DESCRIPTION:
The clinical and research need for noninvasive biomarkers in pulmonary arterial hypertension (PAH) has led the study team to develop 129Xe magnetic resonance imaging (129Xe MRI) to image pulmonary vascular pathology through quantitative 3D maps of gas transfer across the pulmonary blood-gas barrier. 129Xe MRI, in combination with 129Xe spectroscopy (MRS), has a unique signature in PAH and can simultaneously measure capillary blood volume and hemodynamic changes associated with pulmonary vascular remodeling (Wang '19a). This project aims to determine how pulmonary vascular remodeling in PAH at a cellular and pathological level is related to gas exchange physiology changes and hemodynamics (monitored with 129Xe MRI/MRS) and the change in these signals over one year in patients with "stable" PAH. Our central hypothesis is that patients with "stable" PAH will display persistent abnormalities on 129Xe MRI/MRS consistent with pulmonary vascular remodeling and that some patients may have worsening of their disease while appearing to be "stable" disease.

The study team will assess the ability of 129Xe MRI to longitudinally monitor disease progression in patients with "stable" PAH. First, the team will enroll "stable" PAH patients and obtain detailed clinical information to be stored in the REDCAP database. The study team will then follow this cohort of PAH subjects for one year, performing 129Xe MRI scans at baseline, 3 months, 6 months and one year in addition to their standard-of-care assessments including appointments labs, echo, and 6MWTs.

ELIGIBILITY:
Inclusion Criteria:

1. Stable on current treatment regimen and not planning to undergo initiation of new therapy for at least 3 months
2. Outpatients of any gender, Age 18-75
3. WHO functional class (FC) 1-3 symptoms with a diagnosis of group 1 PH (mean pulmonary artery pressures (mPAP) > 20 mmHg, pulmonary capillary wedge pressure (PCWP) ≤ 15mmHg and pulmonary vascular resistance (PVR) ≥3 WU)
4. Willing and able to give informed consent and adhere to visit/protocol schedules (consent must be given before any study procedures are performed).
5. Women of childbearing potential must have a negative urine pregnancy test before MRI

   Exclusion Criteria:
6. Sarcoidosis
7. Active cancer
8. Sickle cell anemia
9. Liver disease (Childs-Pugh class C)
10. Any conditions that prevent the performance of 129Xe MRI scans.
11. Prisoners and pregnant women will not be approached for the study
12. Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine)
13. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary vascular function | Baseline, 3 months, 6 months, 1 year
  Measured by RBC/Membrane metrics on Xe MRI
Change in pulmonary vascular function | Baseline, 3 months, 6 months, 1 year
  Measured by RBC shift metrics on Xe MRI
Change in pulmonary vascular functoin | Baseline, 3 months, 6 months, 1 year
  Measured by RBC amplitude oscillation metrics on Xe MRI

SECONDARY OUTCOMES:
Six Minute Walk Test Distance (6MWD) | Baseline, 3 months, 6 months, 1 year
  Distance patient is able to walk during a six minute walk test
NTproBNP | Baseline, 3 months, 6 months, 1 year
  Lab value of NTproBNP
World Health Organization (WHO) Functional Class (FC) | Baseline, 3 months, 6 months, 1 year
  Change in Functional Class of Pulmonary Hypertension symptoms
Hopsitalizations | Baseline, 3 months, 6 months, 1 year
  Frequency of hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Rajagopal, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No